CLINICAL TRIAL: NCT05154136
Title: A Phase 1, Open-Label, 2-period Drug-Drug Interaction Study to Investigate the Effect of Multiple Doses of Itraconazole on the Single-Dose Pharmacokinetic Profile of AB928 in Healthy Adult Participants
Brief Title: A Drug-Drug Interaction Study to Evaluate the Effect of Itraconazole on the Pharmacokinetic Profile of Etrumadenant in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARC-18
Record Dates: First submitted 2021-10-16; First posted 2021-12-10 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants
Keywords: Etrumadenant; Itraconazole; Healthy participants; Pharmacokinetics; Drug-Drug Interaction; AB928
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Intervention Model Description: The study consists of 2 periods with participants sequentially receiving Treatment A (etrumadenant) in Period 1, followed by Treatment B (etrumadenant + itraconazole) in Period 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etrumadenant then Etrumadenant + Itraconazole (Experimental): Participants will receive the Treatment A (etrumadenant) followed by Treatment B (etrumadenant + itraconazole).
  A washout period of 5 days will be maintained between the two treatments.
  Interventions: Drug: Etrumadenant; Drug: Itraconazole

INTERVENTIONS:
Drug: Etrumadenant — Capsule
  Other Names: AB928
Drug: Itraconazole — Capsule

SUMMARY:
This study will evaluate the effect of multiple oral doses of itraconazole, on the pharmacokinetics of etrumadenant when etrumadenant is administered as a single dose in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female (of non-childbearing potential), at the screening visit
* Body mass index between 18 and 32 kilograms/m^2 inclusive, at screening
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG
* Clinical laboratory test results clinically acceptable at screening and check-in
* Non-smokers or ex-smokers (must have ceased smoking and stopped using nicotine containing products >3 months prior to the first dosing) based on participant self-reporting

Exclusion Criteria:

* Participants who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, rheumatological, endocrine, connective tissue diseases or disorders
* Have a clinically relevant surgical history in the opinion of the principal investigator or designee
* Have a history of relevant atopy or hypersensitivity to the study drugs or related compounds (e.g., allergy to itraconazole or other azole antifungals
* History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing

Note: This is not an exhaustive list of criterias.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Etrumadenant Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
Area Under the Plasma Concentration-time Curve From 0 to Last Observed Non-zero Concentration [AUC(0-t)] of Etrumadenant Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
Area Under the Plasma Concentration Time Curve From Time '0' Extrapolated to Infinity [AUC(0-inf)] of Etrumadenant Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2

SECONDARY OUTCOMES:
Percentage of AUC(0-inf) Extrapolation (AUC%extrap) of Etrumadenant Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
Apparent Total Plasma Clearance (CL/F) of Etrumadenant Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
Time to Cmax (Tmax) of Etrumadenant Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
Apparent First-order Terminal Elimination Rate Constant (Kel) of Etrumadenant Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
Apparent First Order Terminal Elimination Half-life (t1/2) of Etrumadenant Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) of Etrumadenant Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
Cmax of Etrumadenant Metabolites When Etrumadenant is Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
AUC(0-t) of Etrumadenant Metabolites When Etrumadenant is Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
AUC(0-inf) of Etrumadenant Metabolites When Etrumadenant is Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
AUC%extrap of Etrumadenant Metabolites When Etrumadenant is Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
CL/F of Etrumadenant Metabolites When Etrumadenant is Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
Tmax of Etrumadenant Metabolites When Etrumadenant is Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
Kel of Etrumadenant Metabolites When Etrumadenant is Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
t1/2 of Etrumadenant Metabolites When Etrumadenant is Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
Vz/F of Etrumadenant Metabolites When Etrumadenant is Administered With or Without Itraconazole | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Period 1; and Days 5, 6, 7, 9, and 11 during Period 2
Number of Participants with Treatment Emergent Adverse Events | Up to 30 days
  Safety will be assessed by monitoring adverse events and clinically significant changes in 12 lead Electrocardiogram, vital signs, and clinical laboratory tests results.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy